CLINICAL TRIAL: NCT02049372
Title: Developing a Prospective Registry for Complications in Otorhinolaryngologic Surgery: Tonsil Surgery as a Pilot Cohort
Brief Title: Complication Registry for Tonsil Surgery
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Leif Back, MD PhD, University of Helsinki
Other Study IDs: JR/Helsinki/ORL/I
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Tonsillar Surgery Complications
Keywords: complications; tonsillectomy; tonsillotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our aim was to establish a feasible method to prospectively register all tonsil surgery-related complications and to find their possible predictive factors. Our long-term objective is to create a surgical complication registration database, which would provide valuable information for quality assurance and give us a benchmarking tool to improve the results of this surgery in our department.

DETAILED DESCRIPTION:
In a six-month period all patients undergoing tonsillectomy or tonsillotomy with or without adenoidectomy were assessed for enrolment. Demographic and clinical data were recorded prospectively in a database which included 57 variables, such as age, gender, co-morbidities, body mass index, American Society of Anesthesiologists Physical Status Classification, indication for surgery, educational level of surgeon (consultant vs. resident), surgical technique, duration of operation and length of hospital stay.

After the operation, all patients were given instructions to contact our emergency department (ED) if experiencing any adverse event. Incidents of postoperative complications were recorded during the post-surgical visits to the ED. Only complications warranting a visit to the outpatient department or hospital admission were registered.

ELIGIBILITY:
Inclusion Criteria:

* no age limits
* elective tonsillar surgery

Exclusion Criteria:

* procedures carried out due to malignancy
* as a part of multilevel surgery for obstructive sleep apnea
* re-tonsillectomies
* acute operations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: From September 2011 to February 2012, all patients undergoing tonsillectomy or tonsillotomy with or without adenoidectomy were assessed for enrolment.
Sampling Method: Probability Sample
Enrollment: 794 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Complication | September 2011 - February 2012 (6 months)
  After the operation, all patients were given instructions to contact our emergency department (ED) if experiencing any adverse event. Incidents of postoperative complications were recorded during the post-surgical visits to the ED. Only complications warranting a visit to the outpatient department or hospital admission were registered.

SECONDARY OUTCOMES:
Hospital stay | September 2011 - February 2012 (6 months)

OTHER OUTCOMES:
Patient and operative data | September 2011 - February 2012 (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Leif J Bäck, MD PhD, Principal Investigator — Dept of Otorhinolaryngology - Head and Neck Surgery
Locations (1):
- Dept of Otorhinolaryngology - Head and Neck Surgery, Helsinki, Finland

REFERENCES:
- [Derived] Ruohoalho J, Makitie AA, Atula T, Takala A, Keski-Santti H, Aro K, Haapaniemi A, Markkanen-Leppanen M, Back LJ. Developing a Registry for Complications in Otorhinolaryngologic Surgery: Tonsil Surgery as a Pilot Cohort. Otolaryngol Head Neck Surg. 2015 Jul;153(1):34-40. doi: 10.1177/0194599815582156. Epub 2015 Apr 21. PMID 25900187